CLINICAL TRIAL: NCT07145710
Title: Development and Evaluation of Raw Banana Flour-Enriched Muffins for Hypertensive Patients: A Pilot Study
Brief Title: Raw Banana Flour-Enriched Muffins for Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Sana Noreen, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REC-UOL/466/08/24
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-08

CONDITIONS: Hypertension (HTN); Lipid Profile; Liver Enzymes
Keywords: Hypertension; dietary fiber; bioactive compounds; cardiovascular health; functional food; intervention, muffins
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Patients received Whole wheat muffin
  Interventions: Dietary Supplement: Whole wheat muffin enriched with raw banana flour (RBF) (contains 20g RBF)
- 17.5g RBF Group (Experimental): Whole wheat muffin enriched with raw banana flower (RBF) (contains 17.5g RBF)
  Interventions: Dietary Supplement: Whole wheat muffin
- 20 g RBF Group (Experimental): Whole wheat muffin enriched with raw banana flower (RBF) (contains 20g RBF)
  Interventions: Dietary Supplement: Whole wheat muffin enriched with raw banana flour (RBF) (contains 17.5g RBF)

INTERVENTIONS:
Dietary Supplement: Whole wheat muffin — Participants received Whole wheat muffin once a day
  Arms: 17.5g RBF Group
Dietary Supplement: Whole wheat muffin enriched with raw banana flour (RBF) (contains 17.5g RBF) — Participants received Whole wheat muffin enriched with raw banana flour (RBF) (contains 17.5g RBF)
  Arms: 20 g RBF Group
Dietary Supplement: Whole wheat muffin enriched with raw banana flour (RBF) (contains 20g RBF) — Participants received Whole wheat muffin enriched with raw banana flour (RBF) (contains 20g RBF)
  Arms: Placebo group

SUMMARY:
This study evaluated the effects of raw banana flour (RBF)-enriched muffins on hypertensive patients in Lahore, Pakistan. A total of 34 patients were divided into three groups: a control group and two intervention groups receiving muffins with 35% (C1) or 40% (C2) RBF for 10 weeks. Sensory evaluation showed high acceptability of the 35% RBF muffins, comparable to control muffins. Clinical outcomes indicated that both intervention groups experienced improvements in body weight, BMI, blood pressure, liver enzymes, and lipid profiles, with more pronounced benefits observed in the 40% RBF group. The findings suggest that RBF-enriched muffins, particularly at 40% substitution, can offer functional, nutritional, and clinical benefits for individuals with hypertension.

DETAILED DESCRIPTION:
2. Materials and Methods The study received ethical approval from the University of Lahore (REC-UOL/466/08/24). Informed consent was obtained from all participants, who were fully informed about the study's aims, methods, risks, and benefits, and were allowed to ask questions and withdraw at any time.

2.2. Materials Raw banana flour, whole wheat flour, brown sugar, baking powder, pink salt, coconut oil, vanilla essence, cinnamon powder, eggs, and plastic bags were procured from the local market of Lahore, Pakistan, and subsequently stored in the Food Science and Nutrition Lab at the University Institute of Diet and Nutritional Sciences (UIDNS), University of Lahore, Pakistan. Standard kits from Merck Specialities Pvt. Ltd. were employed to assess liver enzyme tests and lipid profiles.

2.3. Settings: This study took place at the Food Science and Nutrition Lab, UIDNS, University of Lahore, and Nutrition Department, Noor Hospital Lahore, Lahore, Pakistan.

2.4. Sensory Evaluation Muffins were tasted by 10 professionals. Randomly placed muffins have two-digit codes. Cookies with two-digit numbers were distributed randomly. The panelists used a 9-point hedonic scale (9 = highly liked; 1 = severely disliked) to rate color, appearance, flavor, texture, overall acceptability, and affordability (Wichchukit & O'Mahony, 2015). During sensory evaluation, panelists cleaned their taste receptors with mineral water and expectorant cups (Handa et al., 2012).

2.5. Subjects In this pilot study, 48 patients signed up; however, 6 of them were not allowed to participate because they did not meet the requirements (Figure 1). We randomly put 42 patients into three groups. There were three groups of 42 patients, each with the same number of people. There were 14 people in each group. Four people were left out of the control group (C0) because of some personal issues. Two people were taken out of the intervention group (C1) because they had to travel, were constipated, or started using an alternative medicine. Two other people moved from the intervention group (C2) to start taking an alternative medicine. Figure 1 shows that 10 patients were in the control group, 12 were in the intervention group (C1), and 12 were in the other intervention group (C2). All of them finished the trial and were tested after 10 weeks, lipid profile and liver enzymes were assessed at the end of study.

2.6 2.9. Statistical analysis All sensory evaluation data were expressed as mean ± standard deviation (SD). One-way analysis of variance (ANOVA) was performed to determine significant differences among the control and raw banana flour-enriched muffin sample groups for each sensory attribute (Steel & Torrie, 1981).

ELIGIBILITY:
Inclusion Criteria:

* The study included men and women between the ages of 35 and 55.
* who had high levels of total cholesterol (>220 mg/dL), total triglycerides (>150 mg/dL), and low-density lipoprotein (>130 mg/dL).

Exclusion Criteria:

* People with diabetes, serious diseases, or surgeries in the last three months, or other conditions that might produce high cholesterol, were not allowed to take part.
* People who had gastrointestinal problems or were known to be allergic to cinnamon were also not accepted.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Lipid Profile | 10 Weeks
  Level of total cholesterol (mg/dL), total triglycerides (mg/dL), and low-density lipoprotein (mg/dL) were measure.
Blood Pressure (systolic pressure and diastolic pressure) | 10 Weeks
  Level of Blood pressure was observed among hypertensive patients

SECONDARY OUTCOMES:
Liver Enzymes | 10 weeks
  Level of Liver function enzymes were observed among participants

CONTACTS AND LOCATIONS:
Locations (1):
- Sana Noreen, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Amini Khoozani A, Kebede B, Birch J, Bekhit AEA. The Effect of Bread Fortification with Whole Green Banana Flour on Its Physicochemical, Nutritional and In Vitro Digestibility. Foods. 2020 Feb 5;9(2):152. doi: 10.3390/foods9020152. PMID 32033343